CLINICAL TRIAL: NCT03784560
Title: Effects of Partial Sleep Deprivation Following Night Shift on Cognitive Functions of Egyptians Anesthesiologists as a Representative of Developing Countries; Prospective Observational Study
Brief Title: Effects of Partial Sleep Deprivation on Cognitive Function of Anesthesiologists
Acronym: sleep
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassant M. Abdelhamid, associate professor, Cairo University
Other Study IDs: N-35-2017
Record Dates: First submitted 2018-12-16; First posted 2018-12-24 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Cognitive Dysfunction; Sleep Deprivation
MeSH Terms: conditions — Cognitive Dysfunction; Sleep Deprivation | interventions — Trail Making Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: anesthesia residents with 24 hours working shift
  Interventions: Other: The Psychomotor Vigilance Task (PVT); Other: Epworth Sleepiness Scale; Other: Karolinska sleeping scale; Other: Trail making test

INTERVENTIONS:
Other: The Psychomotor Vigilance Task (PVT) — PVT has emerged as one of the most widely used tools to assess vigilant attention. Vigilance can be defined as sustained attention and tonic alertness. In sleep deprived individuals, vigilance is the component of cognition that is most consistently and dramatically affected. The PVT is a reaction-time test that allows the collection of a large amount of data in a relatively short period of time. These characteristics increase the sensitivity of the test to detect even small changes in vigilant attention, which can wax and wane within seconds.
  Other Names: PVT
Other: Epworth Sleepiness Scale — Epworth Sleepiness Scale a set of questions that assess excessive daytime sleepiness during professional activities and vacations.
  This scale was designed to assess the efficiency of sleep apnea treatments. It is also used for the subjective sleepiness assessment based on the likelihood of falling asleep in different everyday life situations. This results in an overall score.
  Other Names: ESS
Other: Karolinska sleeping scale — The KSS is assumed to be an ordinal scale with a unitary structure. KSS scores may require standardization to control for differences between subjects. The changes observed in the EEG/EOG with drowsiness do not usually appear until KSS scores reach 7 and higher. Lower KSS scores (<5) may reflect differences in the subjective awareness of fatigue as much, or more than, levels of drowsiness.
  Higher KSS scores (7+) may refer more specifically to the state of drowsiness because the subject may then have experienced involuntary dozing behavior, with "lapsing" episodes and brief loss of awareness of the here-and-now, followed by arousal and the return of awareness, including some awareness of recently having dozed off
  Other Names: KSS
Other: Trail making test — Most variants of this test, which was apparently introduced in 1938 by Partington (Partington & Leiter, 1949), have at least two conditions. In condition A the participant is to draw lines to connect circled numbers in a numerical sequence (i.e., 1-2-3, etc.) as rapidly as possible. In condition B the participant is to draw lines to connect circled numbers and letters in an alternating numeric and alphabetic sequence (i.e., 1-A-2-B, etc.) as rapidly as possible.
  Other Names: TMT

SUMMARY:
The purpose of this study was to evaluate differences in cognitive functions at baseline and following night shift at a trauma center among faculty anesthesiologists.

DETAILED DESCRIPTION:
Anesthesiology is one of the few health-care professions that often demands split-second decisions. This is especially true in a trauma setting where the situation in the operating room can change drastically in a few seconds. Anesthesiologists who cover trauma calls overnight are subject to long work shifts and demanding schedules that may adversely affect their performance. In combination with the disruption of circadian rhythm that can occur with night shift work, decline in performance from the long work shifts can lead to errors in judgment.

An anonymous questionnaire included two groups of different items were used. Items of the first group are about the personal data i.e. age, sex, marital status and parenting status, consumption behavior (tea, coffee, carbonated drinks, tobacco, anxiolytics, antidepressants, psychotropic agents and sport), and professional activity (number of extended worked shifts per month, number of weekends worked per month).

Items of the second group are related to the night shift itself i.e. number of cases, and the rest hours during the shift.

Psychomotor Vigilance Task, Karolinska Sleepiness Scale, Epworth Sleepiness Scale and Trail Making Test before and after the shift were performed.

ELIGIBILITY:
Inclusion Criteria:

* Full-time faculty anesthesiologists employed at Kasr El- Ainy Hospital.
* Both genders
* Ages of 25-28 years.
* Varying levels of experience.

Exclusion Criteria:

* History of chronic neurological disease.
* History of psychiatric disorders such as:

  * Episode of major depression within the past 2 years.
  * Lifetime history of schizophrenia.
  * Other psychotic illness or bipolar illness.

Ages: 25 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: Participants included anesthesiologists employed at Kasr El- Ainy Hospital between the ages of 25-28 years of age and with varying levels of experience.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
The Psychomotor Vigilance Task test | 24 hours
  the participant presses a response button as soon as a visual stimulus appears on the screen. There is standard version of the PVT with duration of 10 min. The shorter version, PVT brief, with duration of 3 minutes have been used in the current study using PEBL 2 software computer program and reaction times (RTs) were displayed to the study participants in milliseconds.

SECONDARY OUTCOMES:
Epworth Sleepiness Scale | at the beginning of the shift, at the end of 24 shift and at the end of the following working day
  the subjects are asked to rate on a scale from 0 to 3 their usual probability of dozing off in 8 different situations, with 0= "would never doze" and 3 = "a high chance of dozing". The total ESS score, ranging from 0 to 24, is the sum score of the eight times. Normal day time sleepiness is represented with scores from 0 to 10 detect, while increased levels of excessive daytime sleepiness are represented with scores of 11-24 represent.
Karolinska sleeping scale | 24 hours
  self-assessed 9-point Likert scale for subjective assessment of the individual's level of drowsiness at a time. It has word descriptors to describe the scale points from 1= "very alert" to 9= "very sleepy, fighting sleep, an effort to keep awake".
Trail making test | 24 hours
  The TMT is formed of two parts. In TMT-A, the subject is asked to draw lines sequentially connecting 25 encircled numbers distributed on a paper sheet. In TMT-B except, the subject is asked to alternate between numbers and letters (e.g., 1, A, 2, B, 3, C, etc.). Each part is represented by time in seconds that required to finish the task.

CONTACTS AND LOCATIONS:
Overall Officials: Bassant abdelhamid, MD, Principal Investigator — Cairo University
Locations (1):
- Anesthesia Department, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided